## Note to File 4

Official Title: A Phase III, Open label, Randomized, Multi-center Study of the Effects of Leukocyte Interleukin, Injection [Multikine] Plus Standard of Care (Surgery + Radiotherapy or Surgery + Concurrent Chemoradiotherapy) in Subjects with Advanced Primary Squamous Cell Carcinoma of the Oral Cavity / Soft Palate Versus Standard of Care Only

NCT Number: NCT01265849

Date: 30 March 2021

March 30, 2021

CEL-SCI Clinical Study CS001P3

Note To File #4

The current SAP Section 7.2 states the following censoring rule. For the ITT population analysis for TCI E, all randomized subjects will be included based on any follow-up post-randomization through study exit. To include all subject follow-up, we will drop this censoring rule.

| Condition | Date of Censoring |
|----------------------------|-------------------|
| Randomized and not treated | Date randomized |

## Signatures:

30 Mar 2021 18:22:035+0000

REASON: I approve this document 5847fe6f-1cee-4c47-ac55-feff592129f2

Yaping Cai

ICON plc

30 Mar 2021 18:37:054+0000

REASON: I have reviewed this document and have no comments that

require addressing. 81797106-ad47-4969-9923-72071d5c68a9

Philip Lavin PhD, FASA, FRAPS Lavin Consulting LLC (CEL-SCI Statistical Consultant) Eyal 7alor Eyal Talor

30 Mar 2021 18:30:059+0000

REASON: I approve this document 5a7c1b19-989b-4b38-8dd9-45225e5fa404

**Eval Talor PhD CEL-SCI Corp** 

John Cipriano John Cipriano 30 Mar 2021 18:25:027+0000

REASON: I approve this document 1ab20719-df7a-48a9-9eff-f62f73358e01

John Cipriano **CEL-SCI Corp**